## The Effect of Education Provided According to Social Cognitive Learning Theory on Diabetes Self - management and Quality of Life in Individuals With Type 2 Diabetes Mellitus

The study was conducted in order to study the effect of the training given according to social cognitive learning theory upon diabetes self-management and quality of life among type 2 diabetes mellitus individuals. The study was done as a randomized-controlled experimental study at Internal Diseases Polyclinics of Afyonkarahisar Public Hospital between November 2021 and August 2022. The study was completed with 60 patients -experimental group (30 patients) and control group (30 patients) who met inclusion criteria. The data were gathered using Information Request Form and Metabolic Variables Form, Diabetes Self-Management Scale (DSMS) for Type 2 Diabetic Patients, Multidimensional Scale of Perceived Social Support (MSPSS), type 2 diabetes mellitus Self-management Questionnaire (SMQ), WHOQOL-BREF (WHO- Quality of Life Scale- Short form). A theoretical and practical training based on social-cognitive learning theory was provided to the experimental group for the first five weeks –one module for each week- through power point presentations and afterwards, SMS reminders were sent every fifteen days for seven weeks and at the end of the twelfth week the training was completed. As for the control group, they received a standard training from diabetes nurse. The data were assessed using suitable statistical methods.

## T.C. AFYONKARAHISAR HEALTH SCIENCES UNIVERSITY CLINICAL RESEARCH ETHICS COMMITTEE DECISIONS

| Meeting Date 03.12.2021 Meeting Number 2021/13 M | Meeting Time | 09:00 | Ethic Committee<br>Code<br>2011-KAEK-2 |
|---|---|---|---|
|---|---|---|---|

569- Dr. Sibel KARACA SiVRİKAYA's application file for Non-Interventional Clinical Studies on "The Effect of Education Given According to Social Cognitive Learning Theory on Diabetes Self-Management and Quality of Life in Individuals with Type 2 Diabetes Mellitus" was reviewed. It was unanimously decided by the members attending the meeting that there was no ethical disapproval in conducting the research, with the responsibility of the researchers, in accordance with the research protocol and taking into account the Ministry of Health's Regulation on Clinical Trials No. 28617 dated 13.04.2013 and the published guidelines.

IT IS LIKE THE ORIGINAL

07.01-2022

Dr. Evrini Sana ARTRAN

Recoorder